CLINICAL TRIAL: NCT02189239
Title: A Phase IV, Randomised, Placebo Controlled Study to Investigate the Effects of Zeller Entspannung Film Coated Tablets on Cortisol Responses in Healthy Volunteers With Acute Stress
Brief Title: Efficacy Study of Zeller Entspannung Film Coated Tablets on Acute Stress
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Max Zeller Soehne AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ze 185-4-2014-02
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: The Primary Condition Studied for This Trial is Acute Stress

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Zeller Entspannung film coated tablets (Active Comparator): Relaxing film coated tablets, 570 mg (Zeller Entspannung Filmtabletten), 3x1 tablet per day for the first three days (morning, midday, evening), at day four 2x1 tablet (morning, midday) preferably during meals with a glass of water.
  Interventions: Drug: Zeller Entspannung film coated tablet
- Placebo tablets (Placebo Comparator): Placebo medication is identical in presentation, color and shape, 3x1 tablet per day for the first three days (morning, midday, evening), at day four 2x1 tablet (morning, midday) during meals with a glass of water.
  Interventions: Drug: Placebo
- No Treatment (Sham Comparator): No medication intake.
  Interventions: Other: No Treatment

INTERVENTIONS:
Drug: Zeller Entspannung film coated tablet
  Arms: Zeller Entspannung film coated tablets
Drug: Placebo
  Arms: Placebo tablets
Other: No Treatment
  Arms: No Treatment

SUMMARY:
The objective of the STRESS trial is to investigate in a mode of action setting the effect of Zeller Entspannung film coated tablets on saliva cortisol response versus Placebo after acute stress in healthy male volunteers. In addition, data on safety and tolerability of Zeller Entspannung will be obtained.

A third arm including no treatment is tested as well. Approximately 72 healthy volunteers will be included into this randomized, double blind study. Study duration will be 7 days, study medication intake will be over 4 days: participants will take the medication one tablet three times a day (morning, midday, evening) the first 3 days, whereas on day 4 only two tablets will be taken (morning and midday).

ELIGIBILITY:
Inclusion Criteria:

* Age:18 - 45 years
* Written informed consent
* Male gender

Exclusion Criteria:

* Any acute or chronic somatic or psychiatric disorder
* Smoking
* Any clinically relevant hepatic disorder
* Any clinically relevant renal disorder
* Any clinically relevant cardiac disorder
* Any clinically relevant respiratory disease (e.g. Asthma)
* Diabetes mellitus
* Any abnormal lab values suggesting diseases from exclusion criteria
* Known allergies to trial medication and excipients
* Alcohol or other drug abuse (e.g. cannabis)
* Concomitant participation in another clinical trial or <4 weeks ago
* Participation in any psychotherapy
* Already participated in a TSST

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The primary objective is to demonstrate in healthy male volunteers that Zeller Entspannung reduces overall saliva cortisol level (AUCg) after acute stress compared with a placebo. | 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Phase I Research Unit, University Hospital Basel, Basel, Switzerland